CLINICAL TRIAL: NCT05540327
Title: A Phase II, Double-blind, Dose-Ranging, Parallel, Long-term Extension Study to Evaluate the Safety and Efficacy of Enpatoran in Participants With Subacute Cutaneous Lupus Erythematosus, Discoid Lupus Erythematosus and/or Systemic Lupus Erythematosus Having Completed the WILLOW (MS200569_0003) Study Treatment (WILLOW LTE)
Brief Title: The Willow LTE Study With M5049 in Participants With SCLE, DLE and/or SLE (WILLOW LTE)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS200569_0048; 2022-000239-21 (EudraCT Number)
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Toll-like Receptor 7; Toll-like Receptor 8; WILLOW; Adults; SLE; CLE; Lupus; Discoid lupus erythematosus; Subacute cutaneous lupus erythematosus; M5049; Enpatoran; LTE
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Erythematosus, Discoid; Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- M5049 low dose + Placebo (Experimental): Participants with CLE (active SCLE and/or DLE) or SLE who received low dose of M5049 in WILLOW study will continue to receive M5049 low dose and matching placebo.
  Interventions: Drug: M5049 low dose; Drug: Placebo
- M5049 medium dose+ Placebo (Experimental): Participants with CLE (active SCLE and/or DLE) or SLE who received medium dose of M5049 in WILLOW study will continue to receive M5049 medium dose and matching placebo.
  Interventions: Drug: M5049 medium dose; Drug: Placebo
- M5049 high dose + Placebo (Experimental): Participants with CLE (active SCLE and/or DLE) or SLE who received M5049 matched placebo or high dose of M5049 in WILLOW study will receive M5049 high dose .
  Interventions: Drug: M5049 high dose; Drug: Placebo

INTERVENTIONS:
Drug: M5049 low dose — Participants will receive film-coated tablets of M5049 at a low dose orally, twice a day (BID) for up to 194 weeks.
  Other Names: Enpatoran
  Arms: M5049 low dose + Placebo
Drug: M5049 medium dose — Participants will receive film-coated tablets of M5049 at a medium dose orally, BID for up to 194 weeks.
  Other Names: Enpatoran
  Arms: M5049 medium dose+ Placebo
Drug: M5049 high dose — Participants will receive film-coated tablets of M5049 at a high dose orally, BID for up to 194 weeks.
  Other Names: Enpatoran
  Arms: M5049 high dose + Placebo
Drug: Placebo — Participants will receive M5049 matching placebo orally, BID for up to 194 weeks.

SUMMARY:
The purpose of the study is to evaluate the long term safety and efficacy of orally administered M5049 in participants with subacute cutaneous lupus erythematosus (SCLE), discoid lupus erythematosus (DLE) and/or systemic lupus erythematosus (SLE) who have completed the 24 week treatment period of Willow study (MS200569_0003 [NCT05162586]).

ELIGIBILITY:
Inclusion Criteria:

* Are SCLE, DLE and/or SLE that have completed the 24 week Treatment of the Willow Study
* Have a Body Mass Index (BMI) within the less than or equal to (<=) 40 kilograms per meter square (inclusive) at Screening
* Participants who had successfully completed Week 48 of the Part 1 will have the opportunity to participate in the LTE Part 2. In exceptional cases and after Sponsor review, participants who have completed the Week 48 visit of the Part 1 within the previous 4-weeks may be considered for Part 2 participation based on eligibility review. Previous 4-weeks will be calculated from the Week 48 visit of Part 1
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants who experienced serious event(s) related to the study intervention during the WILLOW study
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with Long Term Extension (LTE) study participation
* Ongoing or active clinically significant viral (including Severe acute respiratory syndrome coronavirus 2 [(SARS-CoV-2)], bacterial or fungal infection, or any major episode of infection requiring hospitalization
* Received LTE prohibited medication during the WILLOW study or after the WILLOW study Week 24
* Participation in any other investigational drug study after the WILLOW study Week 24
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2028-08-12 (Estimated); Study Completion 2028-08-12 (Estimated)

PRIMARY OUTCOMES:
Part 1: Safety Profile as Assessed by Incidence of Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Adverse Event of Special Interest (AESIs) | Baseline up to Week 50 (Long Term Extension Part 1)
Part 2: Safety Profile as Assessed by Incidence of Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Adverse Event of Special Interest (AESIs) | Baseline up to Week 194 (LTE Part 1 and LTE Prolongation Part 2))

SECONDARY OUTCOMES:
Part 1 and Part 2: Number of Participants with Abnormalities in Laboratory Parameters and QT Interval Corrected | Baseline up to Week 50 and LTE Prolongation up to Week 194 (Part 2)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (122):
- United States (8):
  - The Lundquist Institute at Harbor-UCLA Medical Center, Torrance, California
  - Bay Area Arthritis and Osteoporosis, Brandon, Florida
  - Advance Medical Research Center, Miami, Florida
  - Dawes Fretzin Dermatology Group, LLC, Indianapolis, Indiana
  - AA MRC LLC Ahmed Arif Medical Research Center, Grand Blanc, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Ohio State University - CTMO Parent, Columbus, Ohio
  - Ramesh C Gupta, MD, Memphis, Tennessee
- Argentina (12):
  - Centro de Investigaciones Medicas Mar del Plata - CIM, Buenos Aires
  - CINME - Centro De Investigaciones Metabolicas, Buenos Aires
  - Buenos Aires Skin, Ciudad Autonoma Buenos Aires
  - Hospital Militar Central Dr. Cosme Argerich, Ciudad Autonoma Buenos Aires
  - Centro de Investigaciones Medicas Mar del Plata - CIM, Mar del Plata
  - Instituto de Reumatologia, Mendoza
  - Instituto Medico de alta Complejidad San Isidro S.A (IMAC), San Fernando
  - CER San Juan Centro Polivalente de Asistencia e Inv. Clinica, San Juan
  - Centro Dermatologico Schejtman, San Miguel
  - PSORIAHUE-Medicina Interdisciplinar, San Miguel
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán
- Australia (2):
  - Monash Medical Centre Clayton, Clayton
  - Veracity Clinical Research, Woolloongabba
- Brazil (7):
  - Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte
  - Oncovida - Centro de Onco-Hematologia de Mato Grosso, Cuiabá
  - Clínica SER da Bahia, Graça
  - CMiP - Centro Mineiro de Pesquisa, Juiz de Fora
  - Hospital Moinhos de Vento, Moinhos de Vento
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto - CIP - Centro Integrado de Pesquisa, São José
  - CEPIC - Centro Paulista de Investigação Clínica e Serviços Médicos, São Paulo
- Bulgaria (7):
  - DCC 'Sveti Georgi' EOOD - Cardiology Office, Haskovo
  - MC Artmed OOD, Plovdiv
  - DCC 1 Sevlievo EOOD, Sevlievo
  - DCC Focus 5 - MEOH OOD, Sofia
  - Military Medical Academy - MHAT - Sofia, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD - Clinic of Rheumatology, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD - Clinica of Rheumatology, Sofia
- Chile (6):
  - Clinica Alemana de Osorno - Corporacion de Beneficencia Osorno, Los Lagos
  - BioMedica Research Group - Psicomedica Clinical and Research Group, Santiago
  - CeCim Biocinetic, Santiago
  - Centro Medico Prosalud, Santiago
  - CIEC- Centro Internacional de Estudios Clinicos - Valenzuela Y Compania Ltda, Santiago
  - Dermacross, Santiago
- China (15):
  - The First Affiliated Hospital of Baotou Medical College, Baotou
  - Peking Union Medical College Hospital - Beijing Union Medical College Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Guangdong Provincial People's Hospital, Guangzhou
  - Hainan General Hospital, Haikou
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - The Affiliated Drum Tower Hospital of Nanjing University, Nanjing
  - Huashan Hospital, Fudan University - Neurology, Shanghai
  - Renji Hospital Shanghai Jiaotong University School of Medicine - West Branch, Shanghai
  - Shanghai Skin Disease Hospital, Shanghai
  - West China Hospital, Sichuan University, Sichuan
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
- Colombia (5):
  - Centro de Investigacion Medico Asistencial S.A.S, Barranquilla
  - Centro de Investigacion en Reumatologia y Especialidades Medicas SAS. CIREEM, Bogotá
  - Servimed S.A.S., Bucaramanga
  - Centro Integral de Reumatologia del Caribe SAS CIRCARIBE SAS, Medellín
  - Healthy Medical Center, Zipaquirá
- Greece (2):
  - General Hospital of Athens Laiko, Athens
  - General Hospital Papageorgiou, Thessaloniki
- Chaim Sheba Medical Center - pt, Ramat Gan, Israel
- Japan (9):
  - NHO Asahikawa Medical Center - Dept of Gastroenterology, Asahikawa-shi
  - NHO Chibahigashi National Hospital - Dept of Allergy/Rheumatology, Chiba
  - St. Luke's International Hospital - Dept of Immunology/Allergy, Chūōku
  - Hiroshima University Hospital, Hiroshima
  - Eiraku Clinic - Dept of Rheumatology, Kagoshima
  - Saitama Medical Center - Dept of Rheumatology/Immunology, Kawagoe-shi
  - Kagawa University Hospital - Dept of Immunology/ Rheumatology, Kita-gun
  - Hokkaido University Hospital - Dept of Internal Medicine 2(Rheumatology/Immunolog, Sapporo
  - Tohoku University Hospital - Dept of Hematology/Immunology, Sendai
- CAP Research Ltd, Quatre Bornes, Mauritius
- Mexico (14):
  - Consultorio Privado Dr. Miguel Cortes Hernandez, Cuernavaca
  - Centro de Estudios de Investigacion Basica y Clinica SC, Guadalajara
  - Diseno y Planeacion en Investigacion Medica S.C., Guadalajara
  - Diseño y Planeacion en Investigacion Medica S.C., Guadalajara
  - Centro Medico del Angel, Mexicali
  - CAIMED Investigacion en salud S.A de C.V., Mexico City
  - Clinstile, S.A. de C.V., Mexico City
  - Medical Care & Research SA de CV, Mérida
  - Centro de Investigacion Clínica GRAMEL S.C, México
  - Clinica para el Diagnostico y Tratamiento de las Enfermedades Reumaticas, México
  - Consultorio de Reumatologia - Hospital Angeles Lindavista Cons. 445B, México
  - Grupo Medico Camino S.C., México
  - Centro Regiomontano de Estudios Clínicos Roma S.C., Monterrey
  - CIMAB S.A. de C.V. - Centro de Investigacion Medica Alberto Bazzoni, Torreón
- ICS ARENSIA Exploratory Medicine SRL - Republican Clinical Hospital "Timofei Mosneaga", Chisinau, Moldova
- Philippines (6):
  - Davao Doctors Hospital - Medicine, Davao City
  - Iloilo Doctors Hospital, Iloilo City
  - Mary Mediatrix Medical Center, Lipa City
  - Ospital Ng Makati, Makati City
  - Chinese General Hospital & Medical Center, Manila
  - Far Eastern University - Dr. Nicanor Reyes Medical Foundation - Department of Child Health, Quezon City
- Poland (7):
  - Nova Reuma Domysławska i Rusiłowicz, Spółka Partnerska Lekarza Reumatologa i Fizjoterapeuty, Bialystok
  - Prywatna Praktyka Lekarska prof Pawel Hrycaj, Kościan
  - Centrum Medyczne Plejady, Krakow
  - Centrum Nowoczesnych Terapii Dobry Lekarz, Krakow
  - Twoja Przychodnia PCM, Poznan
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne Sp. z o. o, Szczecin
  - Clinical Best Solutions - Warszawa, Warsaw
- Romania (4):
  - Centrul Medical Monza SRL - Arensia Exploratory Medicine, Bucharest
  - S.C Delta Health Care S.R.L - Ponderas Academic Hospital, Bucharest
  - Spitalul Clinic "Sf. Maria" - Clinica de Medicina Interna si Reumatologie, Bucharest
  - Spitalul Clinic "Sf. Maria" - parent, Bucharest
- Serbia (3):
  - Institute of Rheumatology - Rheumatology, Belgrade
  - Institute of Rheumatology, Belgrade
  - University Clinical Center of Serbia - Clinic of Alergology and Imunology, Belgrade
- South Africa (3):
  - Arthritis Clinical Research Trial Unit - Dr CE Spargo and Dr RB Bhorat, Cape Town
  - University of Pretoria Clinical Research Unit - Parent, Pretoria
  - Naidoo, A - Netcare Umhlanga Hospital, Umhlanga
- South Korea (3):
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Ajou University Hospital, Suwon
- Spain (4):
  - Hospital General de Castellon - Servicio de Reumatologia, Castelló
  - Hospital Regional Universitario de Malaga - Reumatology Dept, Málaga
  - Hospital Universitario Marques de Valdecilla - Servicio de Reumatologia, Santander
  - Hospital Universitario Rio Hortega - Servicio de Medicina Interna, Valladolid
- Taiwan (2):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: https://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200569_0048
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html